CLINICAL TRIAL: NCT03509779
Title: EMT, Reactivation of Embryonic Transcription Factors and Alteration of the miR Signaling Network as Pronostic and Predictive Markers in Lung Cancer
Brief Title: Pronostic and Predictive Value of EMT in Localized Lung Cancer
Acronym: TWISTlung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Georges Pompidou Hospital (Other)
Collaborators: APHP (Other)
Responsible Party: Principal Investigator, Hélène Blons, Professor, European Georges Pompidou Hospital
Other Study IDs: 2013-A01633-42
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: NSCLC, Stage I, II, IIIA, IIIB; Surgery; Progression; Epithelial Mesenchymal Transition
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumor samples analyzed for somatic mutations using NGS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC: NSCLC localized disease treated by surgery

SUMMARY:
The goal of the present research is to identify an "EMT signature", associated with long term disease-free survival after surgery in NSCLC. This study will potentially lead to specific treatment recommendations, thanks to an integrated molecular approach including DNA, RNA and miR profiling In vitro analyses using lung cancer cell lines will subsequently be conducted to validate markers identified in tumor screenings.

DETAILED DESCRIPTION:
One critical issue in studying oncogenesis is the comprehensive understanding of tumor genome complexity. Molecular subtypes may be identified through large-scale molecular screenings or gene expression analyses and molecular signatures are recognized as a relevant source of disease stratification.

The investigators will focus on NSCLC patients with localized diseases included in the ONCOHEGP tissue collection project (OncoHEGP, Ministere de la Recherche n° DC 2009-950). The investigators had previously shown that in EGFR mutated cancer, reactivation of TWIST1 was reversibly linked to EMT and to survival. To go further, the investigators plane to investigate EMT in a large cohort of patients with lung cancer to identify prognostic and predictive markers of long term survival.

The investigators will integrate mutation, and copy number alterations to EMT gene expression analyses and to EMT related miR quantification. Tumor phenotype, miR signatures, mutation status will help classify patients according to survival.

Clinical data will be assessed thanks to the epithor database. Epithor is a government-recognized clinical database, accredited by the French Health Authorities (Haute Autorité de Santé) and is supported by the National Cancer Institute (Institut National du Cancer).

EMT characterization and scoring will be done using 10 markers by qPCR, mutation and CNV screenings by targeted NGS analysis, miRs signature by MIRSeq and qPCR.

ELIGIBILITY:
Inclusion Criteria:

* Patient with NSCLC stage I II IIIA IIIB, treated by surgery at Georges Pompidou Hospital (HEGP) Informed consent ONCOHEGP signed

Exclusion Criteria:

* Informed consent ONCOHEGP not signed

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated by surgery at HEGP having signed the ONCOHEGP consent are eligible to this observational study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-10-20 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival | 1 year
  Time to relapse after surgery
Overall survival | 5 years
  Time to death

SECONDARY OUTCOMES:
Overall survival | 3 years
  Time to death

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Lepimpec Barthes, MD PhD, Principal Investigator — APHP
Locations (1):
- Aphp Hegp, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garinet S, Didelot A, Marisa L, Beinse G, Sroussi M, Le Pimpec-Barthes F, Fabre E, Gibault L, Laurent-Puig P, Mouillet-Richard S, Legras A, Blons H. A novel Chr1-miR-200 driven whole transcriptome signature shapes tumor immune microenvironment and predicts relapse in early-stage lung adenocarcinoma. J Transl Med. 2023 May 15;21(1):324. doi: 10.1186/s12967-023-04086-7. PMID 37189151